CLINICAL TRIAL: NCT00738452
Title: A Phase I Trial of Radioimmunotherapy (Y-90-Mx-DTPA-cT84.66) After Completion of Radiation Therapy Alone, or Radiation Therapy Plus Systemic Therapy in Unresectable or Medically Inoperable, Non-metastatic CEA-Producing Stage I-IIIB Non-Small Cell Lung Cancer
Brief Title: Radiolabeled Monoclonal Antibody Therapy in Treating Patients With Stage I-IIIB Non-Small Cell Lung Cancer After Completion of Radiation Therapy Alone or Combined Radiation Therapy and Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07152; P30CA033572 (NIH); CHNMC-07152; CDR0000611960 (Registry Identifier: NCI PDQ); NCI-2010-01232 (Registry Identifier: NCI CTRP (Clinical Trial Reporting Program)); P01CA043904 (NIH)
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Chromatography, High Pressure Liquid; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemo, monoclonal antibody therapy, radiation) (Experimental): CHEMORADIOTHERAPY: Patients undergo external beam radiation therapy 5 days a week for 45 days. Beginning within 24 hours of the start of radiation therapy, patients receive paclitaxel IV over 1 hour and carboplatin IV over 30 minutes on days 1, 8, 15, 22, 29, and 36 OR cisplatin IV over 60 minutes on days 1, 8, 29, and 36 and etoposide IV over 60 minutes on days 1-5 and 29-33. CONSOLIDATION RADIOIMMUNOTHERAPY: Beginning 6-10 weeks after completion of chemoradiotherapy, patients with stable disease, partial response, or complete response receive a therapeutic dose of yttrium Y 90 anti-CEA monoclonal antibody cT84.66 IV. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: high performance liquid chromatography; Other: pharmacological study; Procedure: radionuclide imaging; Procedure: single photon emission computed tomography; Radiation: radiation therapy; Radiation: yttrium Y 90 anti-CEA monoclonal antibody cT84.66

INTERVENTIONS:
Other: high performance liquid chromatography — Blood evaluation 0 minutes, 1 hour, 4 hours, 1 day, 2 days, 3-5 days and 6-7 days post start of antibody infusion. 24 hour urine sample evaluation daily for 5 consecutive days post antibody infusion.
Other: pharmacological study — Blood evaluation 0 minutes, 1 hour, 4 hours, 1 day, 2 days, 3-5 days and 6-7 days post start of antibody infusion. 24 hour urine sample evaluation daily for 5 consecutive days post antibody infusion.
Procedure: radionuclide imaging — Approximately 1-3 hours, 1 day, 2 days, 3-5 days and 6-7 days post infusion.
Procedure: single photon emission computed tomography — Approximately 2 days and 3-5 days post infusion
Radiation: radiation therapy — 3-6 mCi Indium-111 labeled cT84.66(5mg) and dose escalation (depending on toxicities observed from previous dosages) from a starting dose of 8mCi/m2 Y-90-cT84.66.
Radiation: yttrium Y 90 anti-CEA monoclonal antibody cT84.66 — Dose escalation (depending on toxicities observed from previous dosages) from a starting dose of 8mCi/m2 Y-90-cT84.66.

SUMMARY:
RATIONALE: Radiation therapy uses high energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as carboplatin, paclitaxel, cisplatin, and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiolabeled monoclonal antibodies can find tumor cells and carry tumor-killing substances to them without harming normal cells. Giving radiation therapy and combination chemotherapy together before radiolabeled monoclonal antibody therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of radiolabeled monoclonal antibody therapy when given after radiation therapy and combination chemotherapy in treating patients with stages I-IIIB non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To determine the maximum tolerated dose (MTD) and associated toxicities of intravenous yttrium-90 (90Y) chimeric T84.66 (cT84.66) anti-carcinoembryonic antigen (CEA) antibody targeted radiotherapy delivered after carboplatin/paclitaxel or cisplatin/etoposide and external beam radiotherapy in patients with CEA positive stage III unresectable or medically inoperable non-small cell lung cancer.

SECONDARY OBJECTIVES: I. To collect data on the biodistribution, clearance and metabolism of 90Y (yttrium-90) and 111In (indium-111) chimeric T84.66 administered intravenously. II. To collect data on radiation doses to whole body, normal organs, and tumor through serial nuclear imaging.

OUTLINE: This is a dose-escalation study of yttrium Y 90 anti-CEA monoclonal antibody cT84.66.

CHEMORADIOTHERAPY: Patients undergo external beam radiation therapy 5 days a week for 45 days. Beginning within 24 hours of the start of radiation therapy, patients receive paclitaxel intravenously (IV) over 1 hour and carboplatin IV over 30 minutes on days 1, 8, 15, 22, 29, and 36 OR cisplatin IV over 60 minutes on days 1, 8, 29, and 36 and etoposide IV over 60 minutes on days 1-5 and 29-33.

CONSOLIDATION RADIOIMMUNOTHERAPY: Beginning 6-10 weeks after completion of chemoradiotherapy, patients with stable disease, partial response, or complete response receive a therapeutic dose of yttrium Y 90 anti-CEA monoclonal antibody cT84.66 IV. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for up to 6 months

ELIGIBILITY:
Inclusion criteria:

* Patients must be >= 18 years of age.
* Patients must have a Karnofsky performance status of >= 60%.
* Patients must have histological confirmation non-small cell lung cancer and must have tumors that produce CEA as documented by either immunohistochemistry or by an elevated serum CEA level.
* Patients must have American Joint Committee on Cancer (AJCC) Version 7 Stage I-IIIB non small cell lung cancer (NSCLC) who are not a surgical candidate due to unresectability or medical inoperability.
* Patients must have undergone radiation therapy alone, or radiation therapy plus systemic therapy (which includes chemotherapy or tyrosine kinase inhibitors) as treatment for their lung cancer; patients may receive up to two cycles of consolidative chemotherapy after radiation therapy +/- chemotherapy; this therapy must be completed within 6-12 weeks prior to starting treatment on this trial.
* Patients must have had measurable or evaluable disease prior to receiving standard radiation therapy alone, or radiation therapy plus systemic therapy.
* Patients must have no evidence of progressive disease (therefore, must have stable disease, partial response or complete response) to the therapy given prior to enrollment on this study.
* No radiotherapy, immunotherapy, or chemotherapy within the last 5 years prior to the diagnosis of locally advanced NSCLC; prior adjuvant chemotherapy or tyrosine kinase inhibitor therapy for early stage, resected NSCLC is allowed as long as it was given > 12 months prior to the current diagnosis of locally advanced NSCLC.
* Patients must demonstrate an forced expiratory volume in one second (FEV1) >= 0.9.
* Adequate bone marrow function as evidenced by hemoglobin >= 10 gm %, WBC >= 3500/ul, an absolute granulocyte count of >= 1,500/mm3, and platelets >= 140,000/ul. Patients may be transfused to reach a hemoglobin >=10 gm %.
* Patients must have a total bilirubin <= 1.5 mg/dL and liver transaminases no higher then 2 times the upper limit of normal.
* Patients must have serum creatinine <= 1.5 x upper limit of normal (ULN) and a creatinine clearance >= 45 cc/min (based on Cockcroft Gault formula).
* Patients must not have post-obstructive pneumonia or other serious infection.
* If a patient has previously received murine or chimeric antibody, then serum anti-antibody testing must be negative.
* Serum HIV testing and hepatitis B surface antigen and hepatitis C antibody testing must be negative.
* Women of childbearing potential must have a negative serum pregnancy test prior to entry and while on study must be practicing an effective form of contraception.

Exclusion Criteria:

* Patients with any nonmalignant intercurrent illness (example cardiovascular, pulmonary, or central nervous system disease) which is either poorly controlled with currently available treatment or which is of such severity that the investigators deem it unwise to enter the patient on protocol shall be ineligible.
* Metastatic disease.
* Malignant pleural effusion.
* Patients that did not receive at least 50 Gy thoracic radiation during the course of radiation +/- systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-08-06; Primary Completion 2018-02-07 (Actual); Study Completion 2018-02-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of yttrium Y 90 anti-CEA monoclonal antibody cT84.66 | 6 weeks after treatment
Dose-limiting toxicity | 6 weeks after treatment

SECONDARY OUTCOMES:
Progression-free survival | 6 months after treatment
Overall survival | 6 months after treatment
Sites of recurrence | 6 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Y. Wong, MD, Principal Investigator — City of Hope Comprehensive Cancer Center; Marianna Koczywas, MD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States